CLINICAL TRIAL: NCT03431519
Title: Percutaneous Injection of Strontium Containing Hydroxyapatite Versus Polymethacrylate Plus Short Segment Pedicle Screw Fixation for Traumatic A2 and A3 AO-type Fractures in Adults
Brief Title: Percutaneous Injection Plus Short Segment Pedicle Screw Fixation for Traumatic A2 and A3 AO-type Fractures in Adults
Acronym: NEOGEL
Status: Completed | Type: Observational
Sponsor: University Hospital of Patras (Other)
Collaborators: St. Andrew's General Hospital, Patras, Greece (Other)
Responsible Party: Principal Investigator, Vasileios Syrimpeis, Orthopaedic Surgeon, University Hospital of Patras
Other Study IDs: 2018NEOGEL
Record Dates: First submitted 2018-01-29; First posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Lumbar Fracture; Thoracic Fracture
Keywords: Thoracolumbar fractures; PMMA; KIVA; PEEK
MeSH Terms: conditions — Fractures, Bone | interventions — Vertebroplasty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: The subjects received VP with PEEK and Sr-HA
  Interventions: Procedure: VP
- Group B: The subjects received VP with PEEK and PMMA
  Interventions: Procedure: VP

INTERVENTIONS:
Procedure: VP — Percutaneous Injection of Strontium Containing Hydroxyapatite versus Polymethacrylate plus Short Segment Pedicle Screw Fixation
  Other Names: Vertebroplasty

SUMMARY:
The aim of this study was to examine the short- to medium-term efficacy of percutaneous vertebral body reconstruction by vertebral body augmentation with Sr-HA paste plus short-segment pedicle screw fixation in fresh fractures, as well as to evaluate Sr-HA resorption/substitution. The hypotheses tested in this study were as follows: 1) whether Sr-HA is equivalent to PMMA for restoring the fractured thoracolumbar vertebral body, 2) whether leakage of Sr-HA is less than that of PMMA, and 3) whether Sr-HA is completely resorbed and replaced by cancellous bone.

DETAILED DESCRIPTION:
Introduction Polymethacrylate (PMMA) is commonly used in vertebroplasty and balloon kyphoplasty, but its use has been associated with complications. This study tests three hypotheses: 1) whether strontium hydroxyapatite (Sr-HA) is equivalent to PMMA for restoring thoracolumbar vertebral body fractures, 2) if incidence of PMMA leakage is similar to that of Sr-HA leakage, and 3) whether Sr-HAis resorbed and substituted by new vertebral bone.

Materials and Methods Two age- and sex-matched groups received short percutaneous pedicle screw fixation plus PEEK implant (Kiva, VCF Treatment System, Benvenue Medical, Santa Clara, CA, USA) filled with either Sr-HA (Group A) or PMMA (Group B) after A2- and A3/AO-type thoracolumbar vertebral body fractures. Visual Analog Scale (VAS) score and imaging parameters, which included segmental kyphosis angle (SKA), vertebral body height ratios (VBHr), spinal canal encroachment (SCE), bone cement leakage, and Sr-HA resorption, were compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* One single, severely (>40%) compressed A2 and A3/AO-type thoracolumbar (T10-L3) fracture
* No other serious concomitant injuries

Exclusion Criteria:

* Polytrauma
* Neurologic impairment
* Spinal deformity
* Known malignancy
* Previous fracture or surgery in the same or adjacent vertebrae

Ages: 38 Years to 53 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Female
Study Population: Adult female patients that had a single, severely (>40%) compressed A2 and A3/AO-type thoracolumbar (T10-L3) fracture, without any serious concomitant injuries.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 33 months
  Units on VAS scale (0-10)

SECONDARY OUTCOMES:
Segmental kyphosis angle (SKA) | 33 months
  Angle degrees measured on Xrays
Vertebral body height ratios (VBHr) | 33 months
  Percentage measured on Xrays
Spinal canal encroachment (SCE) | 33 months
  Percentage measured on CT scans
Cement leakage | 33 months
  Yes or no (Boolean value)
Sr-HA resorption | 33 months
  Yes or no (Boolean value)

CONTACTS AND LOCATIONS:
Overall Officials: Vasileios Syrimpeis, MD, Principal Investigator — General Hospital of Patras

IPD SHARING:
Plan to Share IPD: No
Only data published in Scientific Journal Publication

REFERENCES:
- [Derived] Korovessis P, Mpountogianni E, Syrimpeis V, Baikousis A, Tsekouras V. Percutaneous Injection of Strontium Containing Hydroxyapatite versus Polymethacrylate Plus Short-Segment Pedicle Screw Fixation for Traumatic A2- and A3/AO-Type Fractures in Adults. Adv Orthop. 2018 Mar 5;2018:6365472. doi: 10.1155/2018/6365472. eCollection 2018. PMID 29692935